CLINICAL TRIAL: NCT00577135
Title: Diuretic Optimal Strategy Evaluation in Acute Heart Failure (The DOSE-AHF Study)
Brief Title: Determining Optimal Dose and Duration of Diuretic Treatment in People With Acute Heart Failure (The DOSE-AHF Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00017634; U01HL084904-01 (NIH)
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2013-04

CONDITIONS: Heart Failure
Keywords: Loop Diuretics; Furosemide; Fluid Overload; Cardio Renal Failure
MeSH Terms: conditions — Heart Failure; Edema | interventions — Sodium Potassium Chloride Symporter Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Q12 hour bolus (Experimental): Furosemide-Q12 hour bolus
  Interventions: Drug: Furosemide-Low Intensification; Drug: Furosemide-High Intensification
- Continuous Infusion (Experimental): Furosemide-Continuous Infusion
  Interventions: Drug: Furosemide-Low Intensification; Drug: Furosemide-High Intensification
- Low Intensification (Experimental): Furosemide-Low Intensification
  Interventions: Drug: Furosemide-Q12 hour bolus; Drug: Furosemide-Continuous Infusion
- High Intensification (Experimental): Furosemide-High Intensification
  Interventions: Drug: Furosemide-Q12 hour bolus; Drug: Furosemide-Continuous Infusion

INTERVENTIONS:
Drug: Furosemide-Q12 hour bolus — Q12 hours bolus
  Other Names: Loop diuretics
  Arms: High Intensification; Low Intensification
Drug: Furosemide-Continuous Infusion — Continuous infusion
  Other Names: Loop diuretic
  Arms: High Intensification; Low Intensification
Drug: Furosemide-Low Intensification — 1x oral dose
  Other Names: Loop diuretic
  Arms: Continuous Infusion; Q12 hour bolus
Drug: Furosemide-High Intensification — 2.5x oral dose
  Other Names: loop diuretic
  Arms: Continuous Infusion; Q12 hour bolus

SUMMARY:
Heart failure is a disorder in which the heart does not pump blood adequately. This can lead to several serious problems, including reduced blood flow throughout the body, congestion of blood in the veins and lungs, and fluid accumulation in various organs and limbs. Diuretics are often used to address the problem of fluid accumulation, but the optimal dose and the amount of time over which to administer each dose are unclear. This study will compare high and low doses of diuretics administered over longer and shorter periods of time to determine the safest and most effective combination.

DETAILED DESCRIPTION:
Heart failure is a common disorder in which the heart cannot pump enough blood to meet the needs of the rest of the body. Heart failure symptoms include shortness of breath, swelling, and fatigue. Standard treatment for the swelling associated with heart failure includes the use of diuretic medications, such as furosemide, which cause urination and the removal of excess fluids in the body. Although furosemide has been used to treat heart failure patients for many years, it is still unclear how much of the drug to use, and over what time period the drug should be given. This study will evaluate whether furosemide treatment is safer and more effective when the drug is given in high doses versus low doses and in two to three separate doses versus one continuous infusion.

Participants in this study will begin study procedures within the first 24 hours of their hospital admission for heart failure. Participants will be randomly assigned to receive one of the following four treatments: high dose furosemide via continuous intravenous (IV) infusion and placebo every 12 hours via IV bolus; low dose furosemide via continuous IV infusion and placebo every 12 hours via IV bolus; high dose furosemide every 12 hours via IV bolus and placebo via continuous IV infusion; and low dose furosemide every 12 hours via IV bolus and placebo via continuous IV infusion. Each participant will receive treatment for the first 72 hours of his or her hospital stay. Participants will answer questionnaires and undergo physical examinations and blood tests during the first 96 hours of hospitalization and again before hospital discharge or on Day 7, if that occurs first. Participants will be asked to return to their doctors 60 days following hospital discharge to evaluate their responses to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Prior clinical diagnosis of heart failure that was treated with daily oral loop diuretics for at least 1 month
* Current diagnosis of heart failure, as defined by the presence of at least 1 symptom (dyspnea, orthopnea, or edema) AND 1 sign (rales on auscultation, peripheral edema, ascites, pulmonary vascular congestion on chest radiography)
* Daily oral dose of furosemide between 80 mg and 240 mg (or equivalent)
* Identified within 24 hours of hospital admission
* Current treatment plan includes IV loop diuretics for at least 48 hours

Exclusion Criteria:

* Brain natriuretic peptide (BNP) less than 250 mg/mL or N-terminal prohormone brain natriuretic peptide (NT-proBNP) less than 1000 mg/mL
* Received IV vasoactive treatment or ultra-filtration therapy for heart failure since initial presentation
* Treatment plan during current hospitalization includes IV vasoactive treatment or ultra-filtration for heart failure
* Substantial diuretic response to pre-randomization diuretic dosing such that higher doses of diuretics would be medically inadvisable
* Systolic blood pressure less than 90 mm Hg
* Serum creatinine level greater than 3.0 mg/dL at baseline or currently undergoing renal replacement therapy
* Hemodynamically significant arrhythmias
* Acute coronary syndrome within 4 weeks prior to study entry
* Active myocarditis
* Hypertrophic obstructive cardiomyopathy
* Severe stenotic valvular disease
* Restrictive or constrictive cardiomyopathy
* Complex congenital heart disease
* Constrictive pericarditis
* Non-cardiac pulmonary edema
* Clinical evidence of digoxin toxicity
* Need for mechanical hemodynamic support
* Sepsis
* Terminal illness (other than heart failure) with expected survival time of less than 1 year
* History of adverse reaction to the study drugs
* Use of IV iodinated radiocontrast material within 72 hours prior to study entry or planned during hospitalization
* Enrollment or planned enrollment in another randomized clinical trial during this hospitalization
* Inability to comply with planned study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry L. Lee, PhD, Principal Investigator — Duke Clinical Research Institute; Eugene Braunwald, MD, Study Chair — Harvard University
Locations (9):
- United States (8):
  - Morehouse School of Medicine, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Minnesota Heart Failure Network, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Health Sciences Center, Murray, Utah
  - University of Vermont - Fletcher Allen Health Care, Burlington, Vermont
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Result] Felker GM, Lee KL, Bull DA, Redfield MM, Stevenson LW, Goldsmith SR, LeWinter MM, Deswal A, Rouleau JL, Ofili EO, Anstrom KJ, Hernandez AF, McNulty SE, Velazquez EJ, Kfoury AG, Chen HH, Givertz MM, Semigran MJ, Bart BA, Mascette AM, Braunwald E, O'Connor CM; NHLBI Heart Failure Clinical Research Network. Diuretic strategies in patients with acute decompensated heart failure. N Engl J Med. 2011 Mar 3;364(9):797-805. doi: 10.1056/NEJMoa1005419. PMID 21366472
- [Derived] Rasoul D, Zhang J, Farnell E, Tsangarides AA, Chong SC, Fernando R, Zhou C, Ihsan M, Ahmed S, Lwin TS, Bateman J, Hill RA, Lip GY, Sankaranarayanan R. Continuous infusion versus bolus injection of loop diuretics for acute heart failure. Cochrane Database Syst Rev. 2024 May 22;5(5):CD014811. doi: 10.1002/14651858.CD014811.pub2. PMID 38775253
- [Derived] Kelly JP, Cooper LB, Gallup D, Anstrom KJ, Chen HH, Redfield MM, O'Connor CM, Mentz RJ, Hernanadez AF, Felker GM. Implications of Using Different Definitions on Outcomes in Worsening Heart Failure. Circ Heart Fail. 2016 Aug;9(8):e003048. doi: 10.1161/CIRCHEARTFAILURE.116.003048. PMID 27514750
- [Derived] de Denus S, Rouleau JL, Mann DL, Huggins GS, Cappola TP, Shah SH, Keleti J, Zada YF, Provost S, Bardhadi A, Phillips MS, Normand V, Mongrain I, Dube MP. A pharmacogenetic investigation of intravenous furosemide in decompensated heart failure: a meta-analysis of three clinical trials. Pharmacogenomics J. 2017 Mar;17(2):192-200. doi: 10.1038/tpj.2016.4. Epub 2016 Mar 1. PMID 26927285
- [Derived] Lala A, McNulty SE, Mentz RJ, Dunlay SM, Vader JM, AbouEzzeddine OF, DeVore AD, Khazanie P, Redfield MM, Goldsmith SR, Bart BA, Anstrom KJ, Felker GM, Hernandez AF, Stevenson LW. Relief and Recurrence of Congestion During and After Hospitalization for Acute Heart Failure: Insights From Diuretic Optimization Strategy Evaluation in Acute Decompensated Heart Failure (DOSE-AHF) and Cardiorenal Rescue Study in Acute Decompensated Heart Failure (CARESS-HF). Circ Heart Fail. 2015 Jul;8(4):741-8. doi: 10.1161/CIRCHEARTFAILURE.114.001957. Epub 2015 Jun 3. PMID 26041600
- [Derived] Mentz RJ, Stevens SR, DeVore AD, Lala A, Vader JM, AbouEzzeddine OF, Khazanie P, Redfield MM, Stevenson LW, O'Connor CM, Goldsmith SR, Bart BA, Anstrom KJ, Hernandez AF, Braunwald E, Felker GM. Decongestion strategies and renin-angiotensin-aldosterone system activation in acute heart failure. JACC Heart Fail. 2015 Feb;3(2):97-107. doi: 10.1016/j.jchf.2014.09.003. Epub 2014 Oct 31. PMID 25543972
- [Derived] Kociol RD, McNulty SE, Hernandez AF, Lee KL, Redfield MM, Tracy RP, Braunwald E, O'Connor CM, Felker GM; NHLBI Heart Failure Network Steering Committee and Investigators. Markers of decongestion, dyspnea relief, and clinical outcomes among patients hospitalized with acute heart failure. Circ Heart Fail. 2013 Mar;6(2):240-5. doi: 10.1161/CIRCHEARTFAILURE.112.969246. Epub 2012 Dec 18. PMID 23250981
- [Derived] Shah RV, McNulty S, O'Connor CM, Felker GM, Braunwald E, Givertz MM. Effect of admission oral diuretic dose on response to continuous versus bolus intravenous diuretics in acute heart failure: an analysis from diuretic optimization strategies in acute heart failure. Am Heart J. 2012 Dec;164(6):862-8. doi: 10.1016/j.ahj.2012.08.019. Epub 2012 Oct 29. PMID 23194486

RESULTS

PARTICIPANT FLOW:
Groups:
- Q12 Hours Bolus & Low Intensification: Low intensification (1 x oral dose) IV furosemide by Q12 hours bolus
- Q12 Hours Bolus & High Intensification: High intensification (2.5 x oral dose) IV furosemide by Q12 hours bolus
- Continuous Infusion & Low Intensification: Low intensification (1 x oral dose) IV furosemide by continuous infusion
- Continuous Infusion & High Intensification: High intensification (2.5 x oral dose) IV furosemide by continuous infusion
Period: Overall Study
Arm/Group | Q12 Hours Bolus & Low Intensification | Q12 Hours Bolus & High Intensification | Continuous Infusion & Low Intensification | Continuous Infusion & High Intensification
Started | 74 | 82 | 77 | 75
Completed | 74 | 82 | 77 | 75
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Q12 Hours Bolus & Low Intensification | Q12 Hours Bolus & High Intensification | Continuous Infusion & Low Intensification | Continuous Infusion & High Intensification | Total
Number analyzed (Participants) | 74 | 82 | 77 | 75 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (12.4) | 65.2 (13.8) | 64.5 (14.1) | 67.2 (14.0) | 66.0 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 23 | 18 | 82
  Male | 56 | 59 | 54 | 57 | 226

OUTCOME MEASURES:

1. Primary Outcome: Patient Well Being, as Determined by a Visual Analog Scale
Description: Global Visual Analog Scale Scale Range 0-7200; higher score is better
Time Frame: Measured at 72 hours
Population: Each analysis performed for this trial was done twice. The first analysis compared Q12hour versus continuous, the second analysis compared low intensification versus high intensification. The study was not testing the combined 4 way as a pre-specified analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 154 | 149 | 148 | 155
units on a scale | 4236 (1440.4) | 4372.7 (1404.4) | 4170.8 (1436.3) | 4429.6 (1401.4)

2. Primary Outcome: Change in Serum Creatinine
Time Frame: Measured at baseline and 72 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 155 | 146 | 147 | 154
mg/dL | 0.05 (0.30) | 0.07 (0.30) | 0.04 (0.29) | 0.08 (0.31)

3. Secondary Outcome: Change in Weight
Time Frame: baseline and 96 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 151 | 142 | 141 | 152
lbs | -8.0 (7.8) | -9.1 (10.2) | -7.4 (10.1) | -9.6 (7.9)

4. Secondary Outcome: Proportion of Patients Free of Congestion
Time Frame: Measured at 72 hours
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 153 | 144 | 143 | 154
percentage of participants | 14.4 | 15.3 | 11.2 | 18.2

5. Secondary Outcome: Dyspnea, as Determined by Visual Analog Scales
Description: Global Visual Analog Scale Scale Range 0-2400; higher score is better
Time Frame: Measured at 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 153 | 149 | 147 | 155
units on a scale | 1370.8 (486.0) | 1453.8 (518.0) | 1426.0 (504.5) | 1398.2 (502.7)

6. Secondary Outcome: Change in Serum Creatinine
Time Frame: baseline and 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 154 | 146 | 147 | 153
mg/dL | 0.00 (0.18) | 0.01 (0.17) | -0.01 (0.16) | 0.02 (0.19)

7. Secondary Outcome: Change in Cystatin C
Time Frame: baseline and 72 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 125 | 122 | 121 | 126
mg/L | 0.11 (0.30) | 0.17 (0.35) | 0.12 (0.35) | 0.17 (0.31)

8. Secondary Outcome: Change in Serum Creatinine
Time Frame: baseline and 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 155 | 146 | 147 | 154
mg/dL | 0.02 (0.23) | 0.05 (0.26) | 0.01 (0.23) | 0.06 (0.25)

9. Secondary Outcome: Change in Serum Creatinine
Time Frame: baseline and 96 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 155 | 146 | 147 | 154
mg/dL | 0.06 (0.32) | 0.05 (0.32) | 0.05 (0.33) | 0.07 (0.31)

10. Secondary Outcome: Change in Serum Creatinine
Time Frame: baseline and day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 155 | 146 | 147 | 154
mg/dL | 0.10 (0.40) | 0.04 (0.32) | 0.07 (0.33) | 0.08 (0.40)

11. Secondary Outcome: Change in Serum Creatinine
Time Frame: baseline and day 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 117 | 116 | 114 | 119
mg/dL | 0.09 (0.41) | 0.07 (0.45) | 0.09 (0.43) | 0.07 (0.43)

12. Secondary Outcome: Patient Well Being, as Determined by a Visual Analog Scale
Description: Global Visual Analog Scale Scale Range 0-2400; higher score is better
Time Frame: Measured at 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 153 | 149 | 147 | 155
units on a scale | 1280.8 (469.7) | 1303.0 (465.1) | 1288.6 (455.9) | 1294.8 (478.4)

13. Secondary Outcome: Patient Well Being, as Determined by a Visual Analog Scale
Description: Global Visual Analog Scale Scale Range 0-4800; higher score is better
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 153 | 149 | 147 | 155
units on a scale | 2722.6 (940.0) | 2792.6 (932.7) | 2706.5 (931.5) | 2805.2 (939.8)

14. Secondary Outcome: Dyspnea VAS
Description: Dyspnea Visual Analog Scale Scale Range 0-4800; higher score is better
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 153 | 149 | 147 | 155
units on a scale | 2876.6 (960.1) | 3033.1 (1039.3) | 2924.9 (1012.8) | 2981.3 (992.9)

15. Secondary Outcome: Dyspnea VAS
Description: Dyspnea Visual Analog Scale Scale Range 0-7200; higher score is better
Time Frame: 72 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 154 | 149 | 148 | 155
units on a scale | 4455.6 (1468.4) | 4699.1 (1572.7) | 4477.9 (1549.7) | 4668.3 (1496.0)

16. Secondary Outcome: Change in Cystatin C
Time Frame: baseline and day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 137 | 131 | 131 | 137
mg/L | 0.21 (0.43) | 0.16 (0.48) | 0.16 (0.48) | 0.21 (0.42)

17. Secondary Outcome: Change in Cystatin C
Time Frame: baseline and day 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 92 | 98 | 91 | 99
mg/L | 0.20 (0.51) | 0.16 (0.43) | 0.18 (0.47) | 0.18 (0.46)

18. Secondary Outcome: Change in Uric Acid
Time Frame: baseline and 72 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 125 | 121 | 120 | 126
mg/dL | 0.30 (1.02) | 0.44 (1.20) | 0.11 (1.01) | 0.61 (1.15)

19. Secondary Outcome: Change in Uric Acid
Time Frame: baseline and day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 137 | 130 | 130 | 137
mg/dL | 0.40 (1.47) | 0.09 (1.96) | 0.07 (1.69) | 0.42 (1.75)

20. Secondary Outcome: Change in Uric Acid
Time Frame: baseline and Day 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 92 | 99 | 93 | 98
mg/dL | -0.09 (2.28) | -0.71 (2.27) | -0.13 (2.33) | -0.67 (2.24)

21. Secondary Outcome: Change in B-type Natriuretic Peptide
Description: Change in NTproBNP
Time Frame: baseline and 72 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 124 | 121 | 121 | 124
pg/mL | -1316.2 (4364.3) | -1773.2 (3827.5) | -1193.8 (4094.1) | -1881.6 (4105.4)

22. Secondary Outcome: Change in NTproBNP
Time Frame: baseline and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 136 | 130 | 131 | 135
pg/mL | -1133.3 (4883.4) | -1552.0 (4875.8) | -1037.2 (5211.8) | -1629.7 (4524.6)

23. Secondary Outcome: Change in NTproBNP
Time Frame: baseline and Day 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 91 | 98 | 91 | 98
pg/mL | -1449.3 (5010.1) | -1035.1 (6962.9) | -1445.6 (5805.3) | -1038.5 (6364.3)

24. Secondary Outcome: Presence of Cardiorenal Syndrome
Time Frame: Within 72 hours
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 155 | 146 | 147 | 154
percentage of participants | 17.4 | 19.2 | 13.6 | 22.7

25. Secondary Outcome: Treatment Failure
Description: Treatment failure is defined as the patient met cardiorenal syndrome endpoint, worsening or persistent heart failure endpoint, patient died, or there was clinical evidence of overdiuresis requiring intervention within first 72 hours after randomization
Time Frame: Within 72 hours
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 155 | 147 | 147 | 155
percentage of participants | 38.1 | 38.8 | 36.7 | 40.0

26. Secondary Outcome: Net Fluid Loss
Time Frame: Through 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 150 | 140 | 141 | 149
mL | 1595.7 (1476.7) | 1796.4 (1685.1) | 1209.7 (1309.3) | 2149.6 (1681.7)

27. Secondary Outcome: Net Fluid Loss
Time Frame: Through 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 148 | 136 | 139 | 145
mL | 2996.7 (2490.5) | 3120.6 (2504.2) | 2334.8 (2006.4) | 3747.4 (2716.1)

28. Secondary Outcome: Net Fluid Loss
Time Frame: Through 72 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Number analyzed (Participants) | 129 | 113 | 120 | 122
mL | 4236.7 (3207.6) | 4249.2 (3104.3) | 3575.2 (2634.8) | 4898.9 (3478.5)

ADVERSE EVENTS:
Description: Only Serious Adverse Events were collected for this study
Arm/Group | Q 12 Hour Bolus | Continuous Infusion | Low Intensification | High Intensification
Serious Adverse Events (participants affected / at risk) | 69/156 | 67/152 | 76/151 | 60/157
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Q 12 Hour Bolus (N=156) | Continuous Infusion (N=152) | Low Intensification (N=151) | High Intensification (N=157)
Cardiac Failure (Cardiac disorders) | 17 | 18 | 20 | 15
Cardiac Failure Acute (Cardiac disorders) | 13 | 6 | 9 | 10
Ventricular Tachycardia (Cardiac disorders) | 7 | 4 | 7 | 4
Renal Failure (Renal and urinary disorders) | 5 | 6 | 7 | 4
Hypotension (Vascular disorders) | 7 | 9 | 11 | 5
Anemia (Blood and lymphatic system disorders) | 3 | 0 | 2 | 1
Acute Myocardial Infarction (Cardiac disorders) | 4 | 1 | 4 | 1
Cardiac Arrest (Cardiac disorders) | 3 | 3 | 3 | 3
Sepsis (Infections and infestations) | 3 | 4 | 5 | 2
Renal Failure Acute (Renal and urinary disorders) | 3 | 5 | 6 | 2
Angina Pectoris (Cardiac disorders) | 2 | 1 | 2 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 2 | 2 | 1
Atrial Tachycardia (Cardiac disorders) | 1 | 1 | 1 | 1
Cardiac Failure Chronic (Cardiac disorders) | 1 | 3 | 2 | 2
Cardiogenic Shock (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Ventricular Arrhythmia (Cardiac disorders) | 1 | 1 | 2 | 0
Arterial Thrombosis Limb (Vascular disorders) | 1 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 1 | 0
Shock Haemorrhagic (Vascular disorders) | 0 | 1 | 1 | 0
Renal Failure Chronic (Renal and urinary disorders) | 0 | 1 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 2 | 2 | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 6 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No